CLINICAL TRIAL: NCT02723695
Title: Assessment of Perceptual and Postural Performances Following a Cochlear Implantation
Brief Title: Perception and Equilibrium After Cochlear Implantation
Acronym: ORIENTIMPLANT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University of Lorraine (Other)
Responsible Party: Principal Investigator, Cecile PARIETTI-WINKLER, University Professor - Hospital Practitioner, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013-A01086-39
Record Dates: First submitted 2016-03-24; First posted 2016-03-30 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Deafness
Keywords: Cochlear implant; Perception; Posture; Quality of life
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients (Experimental): Surgery (cochlear implantation)
  Interventions: Other: Evaluation of postural performances
- Controls (Active Comparator): Asymptomatic subjects
  Interventions: Other: Evaluation of postural performances

INTERVENTIONS:
Other: Evaluation of postural performances — Postural tests

SUMMARY:
The cochlear implant is an electrical hearing aid that restores the perception of surrounding sounds and speech intelligibility in profoundly deaf patients. During surgery, the labyrinthine break necessary for insertion into the cochlea of the implantable part may cause a malfunction of the vestibular system which can induce dizziness, balance and perception (of the gravitational vertical) disorders. Vestibular compensation and new sonic interactions could alter the balance control and the visual and postural spatial orientation perceptions.

The usual treatment includes the monitoring of the patient's quality of life, of the vestibular function and of hearing. This study adds an assessment of spatial orientation and of posture.

ELIGIBILITY:
Inclusion Criteria:

* Profound deaf patients who are scheduled for a cochlear implantation
* Patients gave their written informed consent
* Patients are affiliated to the french social welfare

Exclusion Criteria:

* Disorders from the motor and/or somesthetic systems (especially the lower limbs)
* Contraindications to the scheduled functional assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-03; Primary Completion 2018-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in postural perception of the gravitational vertical | One year
  The same assessment will be performed 4 times (3 days before surgery, 3 days, 45 days, and one year after surgery).
  The measure is the average difference between the gravitational vertical and the tilt of the platform (in degree) over 20 trials.

SECONDARY OUTCOMES:
Change from baseline in visual perception of the gravitational vertical | One year
  The same assessment will be performed 4 times (3 days before surgery, 3 days, 45 days, and one year after surgery).
  The measure is the average difference between the gravitational vertical and the tilt of the rod (in degree) over 20 trials.
Change from baseline in dynamic balance control | One year
  The same assessment will be performed 4 times (3 days before surgery, 3 days, 45 days, and one year after surgery).
  The composite equilibrium (%) score is calculated over the six conditions of the Sensory Organization Test (Equitest, Neurocom, USA).
Change from baseline in quiet standing within a specific sound environment | One year
  The same assessment will be performed 4 times (3 days before surgery, 3 days, 45 days, and one year after surgery).
  The area covered by the centre of pressure in static posturography (eyes open and eyes closed) is calculated during trials within a specific and controled sound environment [quiet - implant OFF, quiet - implant ON, white noise (70 dB) - implant ON, the semantic content (70 dB) - implant OFF]
Change from baseline in vestibular function | One year
  The same assessment will be performed 4 times (3 days before surgery, 3 days, 45 days, and one year after surgery).
  Vestibular function is quantified by means of videonystagmography (pendular and caloric tests)
Change from baseline in speech recognition | One year
  The same assessment will be performed 4 times (3 days before surgery, 3 days, 45 days, and one year after surgery).
  Speech recognition (in %) is quantified with cochlear phonemic lists of Lafon at 70 dB with and without leep reading.
Change from baseline in quality of life | One year
  The same assessment will be performed 4 times (3 days before surgery, 3 days, 45 days, and one year after surgery).
  Score of the quality of life (QoL) questionnaire (WHOQOL-BREF).
Change from baseline in dizziness | One year
  The same assessment will be performed 4 times (3 days before surgery, 3 days, 45 days, and one year after surgery).
  Self-rated score of the Dizziness Handicap Inventory (DHI).

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Parietti-Winkler, MD, PhD, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- University Hospital of Nancy, Nancy, France